CLINICAL TRIAL: NCT00570531
Title: Phase II Trial of Pre-Operative Chemoradiation Plus Bevacizumab, Followed by Surgery, and Post-Operative Adjuvant Bevacizumab for Patients With Loco-Regional Esophageal Carcinoma
Brief Title: Phase II Trial for Patients With Loco-Regional Esophageal Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was unable the accrue the required number of patients within a reasonable time.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2006.117; HUM 8625 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Loco-regional Esophageal Cancer
MeSH Terms: interventions — Bevacizumab; Paclitaxel; Cisplatin; Fluorouracil; Radiotherapy; Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Experimental)
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel; Drug: Cisplatin; Drug: 5-Fluorouracil; Radiation: Radiation Therapy; Procedure: Esophagectomy

INTERVENTIONS:
Drug: Bevacizumab — Pre-Operative Treatment: Bevacizumab will be given over 60-90 minutes through an I.V. catheter on days # 2 and 16. Post-Operative Treatment:Bevacizumab given over 60-90 minutes through an I.V. catheter every 21 days for 12 months, starting 6-8 weeks after surgery.
  Other Names: Avastin
Drug: Paclitaxel — Pre-Operative Chemotherapy treatment: Paclitaxel 45 mg/m2 will be administered as a 1-hour intravenous infusion on days #2, 9, 16, 23, and 30. It will be given before cisplatin administration.
Drug: Cisplatin — Pre-Operative Chemotherapy Treatment: Cisplatin 30 mg/m2 over 1 hour on days #2, 9, 16, 23, and 30. It will be given after paclitaxel.
Drug: 5-Fluorouracil — Pre-Operative Chemotherapy Treatment: 5-Fluorouracil at 200 mg/m2/day will be given as a continuous intravenous infusion on days #2-33.
Radiation: Radiation Therapy — Pre-Operative Treatment: Radiotherapy will be given Monday through Friday five days a week on days 1-5, 8-12, 15-19, 22-26, and 29-33. Radiotherapy will be administered using MV x-rays. CT scans, the barium swallow, the endoscopy and endoscopic ultrasound reports and PET scans should be used for tumor definition. Post-Operative Radiotherapy: In the event that gross residual disease is left behind at the time of surgery or the patient is found to have a microscopic positive deep or gastric margin following surgery, additional treatment with radiation therapy will be considered.
Procedure: Esophagectomy — Transhiatal esophagectomy performed on approximately Day #57 (6 weeks after last dose of bevacizumab.)

SUMMARY:
The purpose of this study is to determine whether bevacizumab can improve the outcome of treatment for patients with esophageal cancer whose disease is confined to the esophagus or the closely surrounding lymph nodes.

DETAILED DESCRIPTION:
Standard treatment is pre-operative chemotherapy and radiation, followed by surgery. In this study, bevacizumab will be added to the pre-operative chemotherapy and radiation, and then bevacizumab will also be administered for a year after surgery. Bevacizumab is a humanized monoclonal antibody (a type of protein that is normally made by the immune system to help defend the body from infection and cancer) produced by Genentech, Inc. using recombinant DNA technology. Bevacizumab has been approved by the FDA for the treatment of metastatic colorectal cancer in combination with chemotherapy. Bevacizumab is experimental in the treatment of esophageal cancer and has not been approved by the FDA for the treatment of esophageal cancer. Bevacizumab is an antibody directed against vascular endothelial growth factor, or VEGF. VEGF is a growth factor with a well defined role in normal and abnormal blood vessel formation. It is present in a wide variety of normal tissues, but is produced in excess by most solid cancers (tumors). In the setting of cancer, VEGF promotes the growth of blood vessels that bring nutrients to tumor cells. In studies with laboratory animals, bevacizumab inhibits the growth of several different types of human cancer cells, including colon cancer cells, by blocking the effects of VEGF. By blocking VEGF, your doctors hope that bevacizumab may decrease blood supply to the tumor, and therefore decrease the ability of the tumor to grow and come back after chemotherapy, radiation, and surgery.

ELIGIBILITY:
Inclusion Criteria:

1. No prior treatment for esophageal cancer
2. No prior radiation to the chest or upper abdominal area
3. No prior treatment with an EGFR inhibitor or an anti-angiogenic agent
4. Disease should be limited to the esophagus and regional lymph nodes -

Exclusion Criteria:

1. History of stroke
2. History of heart attack
3. Inadequately controlled high blood pressure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-06; Primary Completion 2010-10 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Urba, MD, Principal Investigator — University of Michigan Rogel Cancer Center

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab: Bevacizumab: Pre-Operative Treatment: Bevacizumab will be given over 60-90 minutes through an I.V. catheter on days 2 and 16. Post-Operative Treatment:Bevacizumab given over 60-90 minutes through an I.V. catheter every 21 days for 12 months, starting 6-8 weeks after surgery.
  Paclitaxel: Pre-Operative Chemotherapy treatment: Paclitaxel 45 mg/m^2 will be administered as a 1-hour intravenous infusion on days 2, 9, 16, 23, and 30. It will be given before cisplatin administration.
  Cisplatin: Pre-Operative Chemotherapy Treatment: Cisplatin 30 mg/m^2 over 1 hour on days 2, 9, 16, 23, and 30. It will be given after paclitaxel.
  5-Fluorouracil: Pre-Operative Chemotherapy Treatment: 5-Fluorouracil at 200 mg/m2/day will be given as a continuous intravenous infusion on days #2-33.
  Radiation Therapy: Pre-Operative Treatment: Radiotherapy will be given Monday through Friday five days a week on days 1-5, 8-12, 15-19, 22-26, and 29-33. Radiotherapy will be administered using MV x-rays.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 60 [44 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival Time
Description: The primary outcome that will be measured is the length of time that patients are alive without recurrence of cancer following this therapy.
Time Frame: 5 years
Population: The study was unable to accrue the number of patients necessary to analyze the primary objective.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 0

2. Secondary Outcome: The Number of Patients Cancer Free at the Time of Surgery
Description: Determination of whether the pre-operative treatment can eliminate all the cancer cells at the time of surgery.
Time Frame: 1 year
Population: The study was unable to accrue the number of patients necessary to analyze the objective.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 0

3. Secondary Outcome: The Proportion of Toxicities Experienced by Participants
Description: To assess the toxicity of this regimen.
Time Frame: Every three weeks for one year
Population: The study was unable to accrue the number of patients necessary to analyze the objective.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=6)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 1 (2)
Weight loss (Investigations) | 1 (1)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Leak (including anastomotic), GI (Gastrointestinal disorders) | 1 (1)
Necrosis, GI (Gastrointestinal disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hemorrhage, GI (Vascular disorders) | 1 (1)
Infection (Lung) (Infections and infestations) | 1 (1)
Infection (Mediastinum) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (2)
Fistula, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=6)
Allergic Rhinitis (Immune system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 4 (11)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (4)
Lymphopenia (Blood and lymphatic system disorders) | 2 (6)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Prolonged QTc interval (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (4)
Atrial flutter (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Cardiopulmonary arrest, cause unknown (non-fatal) (Cardiac disorders) | 1 (3)
Hypertension (Cardiac disorders) | 1 (2)
Hypotension (Cardiac disorders) | 2 (2)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (6)
Fever (in the absence of neutropenia) (General disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (2)
Rigors/chills (General disorders) | 2 (2)
Weight loss (Investigations) | 6 (12)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 1 (2)
Anorexia (Gastrointestinal disorders) | 3 (5)
Constipation (Gastrointestinal disorders) | 3 (3)
Dehydration (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 5 (8)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 4 (9)
Esophagitis (Gastrointestinal disorders) | 3 (3)
Fistula, GI (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 2 (2)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
Ileus, GI (functional obstruction of bowel) (Gastrointestinal disorders) | 1 (1)
Leak (including anastomotic), GI (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 4 (4)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (11)
Necrosis, GI (Gastrointestinal disorders) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2 (6)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hemorrhage, GI (Vascular disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory (Vascular disorders) | 2 (2)
Colitis, infectious (Infections and infestations) | 1 (1)
Infection (Lung) (Infections and infestations) | 1 (1)
Infection with Grade 3 or 4 neutrophils (Mediastinum) (Infections and infestations) | 1 (1)
Infection with normal ANC (Mediastinum) (Infections and infestations) | 1 (3)
Infection with normal ANC (Sinus) (Infections and infestations) | 1 (1)
Infection with normal (Upper Aerodigestive) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (2)
Edema: limb (General disorders) | 2 (2)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (6)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 2 (5)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (6)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2 (12)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (4)
Joint-function (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Dizziness (Nervous system disorders) | 1 (2)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Mood alteration (Nervous system disorders) | 2 (2)
Mood alteration (Nervous system disorders) | 3 (3)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Pain, Abdomen (Gastrointestinal disorders) | 3 (3)
Pain, Back (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain, Eosphagus (Gastrointestinal disorders) | 2 (3)
Pain, Head (Nervous system disorders) | 1 (1)
Pain, Joint (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain, Muscle (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Neck (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain, Oral Cavity (Gastrointestinal disorders) | 1 (1)
Pain, NOS (General disorders) | 1 (2)
Pain, Throat (Gastrointestinal disorders) | 2 (2)
Pain - Other (General disorders) | 1 (2)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fistula, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 3 (3)
Vascular - Other (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was unable the accrue the required number of patients within a reasonable time and therefore the primary objective was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes